CLINICAL TRIAL: NCT00559624
Title: A Phase I/II Open Label Dose Escalation Study to Investigate the Safety and Tolerability of Acadesine in Patients With B-cell Chronic Lymphocytic Leukemia
Brief Title: Safety and Tolerability Open Label Dose Escalation Study of Acadesine in B-CLL Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advancell - Advanced In Vitro Cell Technologies, S.A. (Industry)
Collaborators: Nexus Oncology Ltd (Unknown)
Responsible Party: Clara Campàs i Moya, PhD, Advancell - Advanced In Vitro Cell Technologies, S.A.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATH001-CLN01
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Leukemia, B-Cell, Chronic
Keywords: safety; tolerability; dose-escalation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acadesine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Acadesine — For part I of the study one 4 hour intravenous infusion will be given. In part II upto five 4 hour intravenous infusions will be given over 20 days.
  Other Names: Acadra

SUMMARY:
The main aim of this study is to test the safety of acadesine in patients with B-CLL and see what effects it has on patients and their leukaemia. The study also aims to examine the way acadesine is processed by the body. The study will look at the effects of acadesine in the body and the concentration of the drug and its main by-product (ZMP) in the blood to determine the dose and the frequency of dosing that is likely to be the most effective.

DETAILED DESCRIPTION:
This is a Phase I/II, open-label, escalating dose and number of doses study that will involve up to 30-40 patients with B-CLL. A patient who fails to reach their final assessment visit due to reasons other than the occurrence of a dose limiting toxicity (DLT) may be replaced. Eligible patients will be enrolled into Part I or Part II of the study in cohorts of three patients. There will be a requirement to stagger Day 1 dosing between all patients in each cohort by a minimum of 48 hours. In the first part of the study (Part I) patients will receive a single dose of acadesine on Day 1. In the second part of the study (Part II), patients will receive up to 5 doses of treatment over a period of up to 20 days starting on Day 1.

In Part I of the study, the starting dose will be 50 mg/kg given as a 4 hour iv infusion on Day 1 only. Patients will continue to be assessed for safety, pharmacokinetics (PK) and pharmacodynamics for up to three weeks after dosing (to Day 22). The decision to escalate to the next dose in a separate cohort of patients will be based on the assessment of safety, including any DLTs, pharmacokinetic modelling (PKM) of exposure to ZMP and pharmacodynamic response data, where available, by an independent Data Monitoring Board (DMB). A DLT is defined as a Grade 3 or 4 toxicity, which may be local to the injection site or systemic, which is observed within 21 days of dosing and is considered to be related to study drug. The dose will not be escalated if PKM indicates that the exposure to ZMP has reached a plateau.

Dose escalation will continue with each new cohort in accordance with the rules described in the following table. The dose below that at which dose escalation is stopped will be considered the Optimal Biological Dose (OBD) and this dose will be the starting dose used in Part II of the study which will assess repeat dosing with acadesine. The OBD will be reviewed by the DMB prior to the start of Part II of the study.

If a DLT is noted in a given cohort in Part I, the following dose escalation rules will be followed to ascertain the maximum administered dose (MAD). In the unlikely event that a DLT is seen in ≥ 2 patients at the starting dose used in Part I, the study may be resumed with a lower dose if there is adequate evidence of the desired pharmacodynamic effect, ie a reduction in B-cell count, at the starting dose.

Dose escalation in Part I of the study shall follow a modified Fibonacci dose escalation design, with 100% dose escalations allowed until a Grade 2 toxicity that is considered related to treatment is confirmed (as defined by the NCI CTCAE v3.0). If this occurs, future escalations shall then be incremental (67%, 50%, 40%, 33%, etc), until the MAD is confirmed. Intermediate dose levels may be evaluated if indicated by the acquired safety or PK data.

In Part I of the study, blood samples for PK analysis (for both acadesine and its metabolite ZMP) will be taken pre-dose and 0, 30, 60 minutes, 2, 6, 20, 72, 96, and 168 hours, 14 and 21 days post-dose in all cohorts. Predictive modelling of repeat dose pharmacokinetics will be carried out and used in conjunction with the safety and pharmacodynamic data to predict a suitable multiple dose regimen in Part II of the clinical study, where up to 5 doses will be administered at regular intervals over a period of up to 20 days. The Part II dosing decision will be based on a review of the data by the DMB.

In Part II one additional acadesine dose will be administered for each successive new cohort enrolled. The decision to add an additional dose in a separate cohort of patients will be based on assessment of safety, including any DLTs, PKM of exposure to ZMP, and pharmacodynamic response data, where available, by the DMB. Blood samples for PK analysis in Part II of the study will be taken pre-dose and at 0, 30, 60 minutes, 2, 6, 20, 72, 96, and 168 hours post-dose on the first and last day of dosing and also at pre-dose and 0 minutes post-dose for any interim doses. Samples will also be taken 14 and 21 days after completion of the last dose for each patient.

As in Part I, patients in Part II will continue to be followed up for 21 days after their last dose of acadesine. If 1 out of the 3 patients experiences a DLT, a further 3 patients will be recruited to the cohort. If ≥ 2 patients out of the 6 experience a DLT, dosing will be stopped for this cohort and further cohorts of patients may be enrolled to receive up to 5 administrations of acadesine at a lower dose (or intermediate dose) over a 20 day period, based on safety, pharmacodynamic and pharmacokinetic data. The decision to continue at a lower dose will be based on a review by the DMB.

Sampling times for pharmacokinetic assessments may be altered during the study based on the data collected in order to fully define the pharmacokinetic profile of acadesine and ZMP. The total volume of blood required for these assessments will not increase.

ELIGIBILITY:
Inclusion Criteria:

* B-CLL patients with refractory or relapsed disease who have received one or more (≥ 1) prior lines of treatment which must have included either a fludarabine based regimen or an alkylator based regimen. Refractoriness is defined as any patient who has failed to achieve a CR, nPR or PR according to the National Cancer Institute (NCI) working group guidelines for CLL. Fludarabine refractoriness will also include patients who achieved a CR, nPR or PR of ≤ 6 months duration.
* Diagnosis of B-CLL according to NCI Working Group Criteria.
* Have an elevated B-cell count of ≥ 5000/mm3.
* Have a T-cell count ≥ 200/mm3.
* ECOG Performance Status ≤ 2.
* Have a life expectancy of at least 3 months.
* Age ≥ 18 years, of either gender.
* Have given written informed consent, prior to any study related procedure not part of the patient's normal medical care
* Receive allopurinol prophylaxis for hyperuricaemia.

Exclusion Criteria:

* Patients who, in the opinion of the Investigator, need immediate treatment with proven chemotherapy and/or immunotherapy, and/or transplantation.
* Have B-CLL with central nervous system involvement.
* Have participated in any other investigational drug study or have undergone an experimental therapeutic procedure considered to potentially interfere with the study in the 30 days preceding Day 1.
* Have received chemotherapy or radiotherapy treatment in the 30 days preceding Day 1.
* Require oral or parenteral steroids with the exception of inhaled steroids or low-dose oral steroids (<10mg prednisolone per day or equivalent) for an indication other than B-CLL.
* Have a serious medical or psychiatric condition that could, in the Investigator's opinion, potentially interfere with their treatment and/or participation in the study.
* Have uncontrolled diabetes mellitus
* Have a history of gout.
* Have a serious concomitant disease including:

  * Significant cardiac disease - New York Heart Association Classes III or IV or have suffered a myocardial infarction in the last 6 months.
  * Chronic pulmonary obstructive disease with hypoxemia.
  * Clinically active auto-immune disease.
  * Active infection such as tuberculosis, CMV (Cytomegalovirus).
* Any secondary malignancy requiring active treatment (except hormonal therapy).
* Have inadequate bone marrow reserve: neutrophils < 1.0 x 109/L, platelet count < 50 x 109/L (unsupported by transfusion), or coagulation abnormalities.
* Have inadequate liver function: total bilirubin > 1.5 x upper limit of normal values (ULN), AST, ALT, or alkaline phosphatase > 2.5 x ULN.
* Have inadequate renal function, defined by serum creatinine ≥ 1.5 x ULN, unless creatinine clearance is measured and found to be at least 60 mL/min.
* Have serum uric acid levels outside the normal range.
* Females of childbearing potential who are unwilling to employ adequate means of contraception (hormonal contraceptive, intrauterine device, diaphragm with spermicide or condom with spermicide) for the duration of the study and 30 days after the last acadesine administration.
* Pregnant or lactating females.
* Male patients who are not surgically sterile and who are unwilling to use a condom with spermicide for the duration of the study and for 3 months after the last acadesine administration.
* Abuse of alcohol or other recreational drugs.
* Known HIV or Hepatitis B (unless clearly due to vaccination) or C positive.
* Known allergy to acadesine or any of its excipients.
* Have undergone previous allogeneic stem cell transplant.
* Transformation to Richter's syndrome or other aggressive B-cell malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
adverse event and serious adverse events(incidence, causality, severity), local tolerability (including liver enzymes, blood glucose and uric acid) and vital signs. | up to and including Day 22 follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Den Neste, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (8):
- Belgium (3):
  - Hematology Department, ZNA Stuivenberg, Antwerp
  - Cliniques universitaires Saint-Luc Haematology Dept, Brussels
  - Hematology Department UZ Gasthuisberg, Leuven
- France (2):
  - Hôpital Avicenne, Bobigny
  - Service des maladies du sang Hôpital HURIEZ, CHRU, Lille
- Spain (3):
  - Hematologia Clinica, Institut Catala d'Oncologia, Barcelona
  - Hospital Madrid Nortesanchinarro, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia